CLINICAL TRIAL: NCT05633147
Title: Effect of Repeated Dosing of Clarithromycin on PK of Linaprazan Glurate/Linaprazan, Effect of Single Dose of Linaprazan Glurate on PK of Clarithromycin, Single/Repeated Dosing of Linaprazan Glurate on PK of Midazolam to Healthy Subjects
Brief Title: Effect of Clarithromycin on PK of Linaprazan, Linaprazan on PK of Clarithromycin and Linaprazan on PK of Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cinclus Pharma Holding AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CX842A2105
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Safety Issues; Pharmacokinetics; Drug Interaction; Tolerability
MeSH Terms: interventions — Drug Interactions; Didanosine; Clarithromycin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- linaprazan glurate (Experimental): Part I: Linaprazan glurate in base form, 100 mg once daily will be administered under fasting conditions at day 1 and day 10.
  Part II: Linaprazan glurate hydrochloride (HCl), 75 mg twice a day for 13 days. The morning dose will be administered under fasting conditions on Day 2 and Day 14.
  Interventions: Drug: Linaprazan glurate; Drug: Drug drug interaction (DDI) - Clarithromycin (Part I); Drug: Drug drug interaction (DDI) - Midazolam (Part 2)

INTERVENTIONS:
Drug: Linaprazan glurate — Investigational Medicinal Product: Linaprazan glurate (tablets).
  Part I:
  Linaprazan glurate in base form, 100 mg once daily Day 1 and Day 10.
  Part II:
  Linaprazan glurate hydrochloride (HCl), 75 mg twice daily for 13 days.
Drug: Drug drug interaction (DDI) - Clarithromycin (Part I) — Index inhibitor (perpetrator drug) Clarithromycin 500 mg twice daily for 9 days (tablets).
Drug: Drug drug interaction (DDI) - Midazolam (Part 2) — Substrate for CYP3A. Midazolam 2.5 mg once daily (2.5 mL oral solution).

SUMMARY:
This is a phase I, open-label, fixed sequence design, drug-drug-interaction (DDI) study divided in 2 parts. Part I is designed to evaluate whether concomitant treatment with linaprazan glurate and clarithromycin, a strong inhibitor of cytochrome P450 3A4 (CYP3A4) and P-glycoprotein P (PgP), leads to an effect on the systemic exposure to linaprazan glurate and linaprazan and whether there is an effect on the pharmacokinetics of clarithromycin after a single dose of linaprazan glurate. Part II is designed to evaluate the effect of repeated doses of linaprazan glurate on the pharmacokinetics (PK) of a sensitive substrate of CYP3A (midazolam).

ELIGIBILITY:
Main Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male and female subjects of non-childbearing potential aged 18 to 60 years, inclusive.
3. Body mass index ≥ 18.0 and ≤ 30.0 kg/m2.
4. Subjects as well as their partners, must agree to contraception requirements. Male subjects must refrain from donating sperm.

Main Exclusion Criteria:

1. Have known allergies to any components of the linaprazan glurate formulation, to clarithromycin/midazolam or to any drugs of a similar class including excipients associated with any of the drugs.
2. Use of CYP3A4 inhibitors, antacids, PPIs or any medication that changes gastric pH.
3. Use of any prescribed or non-prescribed CYP3A4-inducing medication or other metabolic enzyme inducers.
4. History of any clinically significant disease or disorder defined in the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-11-27 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Palm, Study Director — CTC Clinical Trial Consultants AB
Locations (1):
- CTC Clinical Trials Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from CTC's database of volunteers and from advertising in media (including social media).
Pre-assignment Details: Screening details:
  The screening visits were performed within 28 days prior to dosing (Day 28 to Day -1) for both parts.
  Part I: 27 subjects were screened and 17 subjects were included in Part I of the study.
  Part II: 56 subjects were screened and 18 subjects were included in Part II of the study.
Groups:
- Period I, Part I: Linaprazan glurate in base form, tablets 100 mg administered under fasting conditions Day 1 and Day 10.
  Drug drug interaction (DDI) - Clarithromycin (Part I): Index inhibitor (perpetrator drug) Clarithromycin 500 mg twice daily for 9 days (tablets).
- Period II, Part II: IMP Linaprazan glurate hydrochloride (HCl), tablets 75 mg twice daily for 13 days. Morning dose administered under fasting conditions on Day 2 and Day 14.
  Drug drug interaction (DDI) - Midazolam: Substrate for CYP3A. Midazolam 2.5 mg once daily (2.5 mL oral solution) Day 1, Day 2 and Day 14.
Period: Overall Study
Arm/Group | Period I, Part I | Period II, Part II
Started | 17 | 18
Completed | 16 | 18
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I: Linaprazan glurate in base form, tablets 100 mg administered under fasting conditions Day 1 and Day 10.
  Drug drug interaction (DDI) - Clarithromycin (Part I): Index inhibitor (perpetrator drug) Clarithromycin 500 mg twice daily for 9 days (tablets).
- Part II: IMP Linaprazan glurate hydrochloride (HCl), tablets 75 mg twice daily for 13 days. Morning dose administered under fasting conditions on Day 2 and Day 14.
  Drug drug interaction (DDI) - Midazolam: Substrate for CYP3A. Midazolam 2.5 mg once daily (2.5 mL oral solution) Day 1, Day 2 and Day 14.
- Total: Total of all reporting groups
Arm/Group | Part I | Part II | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (13.0) | 35.0 (12.3) | 36.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Period I, Part I - Linaprazan Glurate and Linaprazan PK Parameters With and Without Co-administration of Clarithromycin - AUC0-inf
Description: Area under the plasma concentration curve from 0 to infinity (AUC0-inf). The AUC were calculated to the time point of the last quantifiable plasma concentration and then extrapolated to infinity using the concentration in the last quantifiable sample and the estimated terminal elimination rate constant (Lambdaz).
Time Frame: Timepoints collected: pre-dose, 15 min, 30 min, 45 min, 1.15 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 18 h, 24 h, 36 h, 48 h and 72 h after dosing (on dosing Days 1 and 10).
Population: Data is presented for:
  * Linaprazan (active metabolite) after 100 mg single dose administered alone
  * Linaprazan (active metabolite) after 100 mg single dose co-administered with clarithromycin
  * Linaprazan glurate (prodrug) after 100 mg single dose administered alone
  * Linaprazan glurate (prodrug) after 100 mg single dose co-administered with clarithromycin
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Part I
Number analyzed (Participants) | 16
h*nmol/L
  Linaprazan (alone) | 13950 (5649)
  Linaprazan (co-admin) | 42840 (16260)
  Linaprazan glurate (alone) | 137.3 (52.02)
  Linaprazan glurate (co-admin) | 165.9 (79.56)

2. Primary Outcome: Period I, Part I - Linaprazan Glurate and Linaprazan PK Parameters With and Without Co-administration of Clarithromycin - AUC0-t
Description: AUC from time 0 to time t (AUC0-t). AUC0-t were analyzed using a mixed model following a natural logarithmic transformation, with fixed effect for treatment and random effect for subject.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Part I
Number analyzed (Participants) | 16
h*nmol/L
  Linaprazan (alone) | 13870 (5346)
  Linaprazan (co-admin) | 39870 (13840)
  Linaprazan glurate (alone) | 133.6 (51.87)
  Linaprazan glurate (co-admin) | 160.6 (81.64)

3. Primary Outcome: Period I, Part I - Linaprazan Glurate and Linaprazan PK Parameters With and Without Co-administration of Clarithromycin - Cmax
Description: Maximum plasma concentration (Cmax). Cmax were analyzed using a mixed model following a natural logarithmic transformation, with fixed effect for treatment and random effect for subject.
Time Frame: and 72 h after dosing (on dosing Days 1 and 10).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part I
Number analyzed (Participants) | 16
nmol/L
  Linaprazan (alone) | 1844 (712.4)
  Linaprazan (co-admin) | 2742 (1217)
  Linaprazan glurate (alone) | 131.1 (53.72)
  Linaprazan glurate (co-admin) | 176.8 (114.3)

4. Primary Outcome: Period II, Part II- Midazolam PK Parameters in the Presence and Absence of Linaprazan Glurate Administration - AUC0-inf
Description: Area under the plasma concentration curve from 0 to infinity - AUCinf. AUC were calculated to the time point of the last quantifiable plasma concentration and then extrapolated to infinity using the concentration in the last quantifiable sample and the estimated terminal elimination rate constant (Lambdaz).
Time Frame: Timepoints collected: Pre-dose, 15 min, 30 min, 1 h, 2 h, 4 h, 8 h, 12 h, 14 h, 20 h and 24 h (on day 1, 2 and 14).
Population: Data is presented for:
  * Midazolam alone, Day 1
  * Midazolam co-administered with linaprazan glurate, Day 2
  * Midazolam co-administered with linaprazan glurate, Day 14
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part II
Number analyzed (Participants) | 17
h*ng/mL
  Midazolam (alone) | 38.57 (13.98)
  Midazolam (co-admin) Day 2 | 40.78 (16.04)
  Midazolam (co-admin) Day 14 | 33.06 (10.46)

5. Primary Outcome: Period II, Part II- Midazolam PK Parameters in the Presence and Absence of Linaprazan Glurate Administration - AUC0-t
Description: AUC from time 0 to time t - AUC0-t. AUC0-t were analyzed using a mixed model following a natural logarithmic transformation, with fixed effect for treatment and random effect for subject.
Time Frame: Timepoints collected: Pre-dose, 15 min, 30 min, 1 h, 2 h, 4 h, 8 h, 12 h, 14 h, 20 h and 24 h (on day 1, 2 and 14).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part II
Number analyzed (Participants) | 17
h*ng/mL
  Midazolam (alone) | 37.12 (13.86)
  Midazolam (co-admin) Day 2 | 39.66 (16.01)
  Midazolam (co-admin) Day 14 | 32.19 (10.41)

6. Primary Outcome: Period II, Part II- Midazolam PK Parameters in the Presence and Absence of Linaprazan Glurate - Cmax
Description: Maximum plasma concentration - Cmax. Cmax were analyzed using a mixed model following a natural logarithmic transformation, with fixed effect for treatment and random effect for subject.
Time Frame: Timepoints collected: Pre-dose, 15 min, 30 min, 1 h, 2 h, 4 h, 8 h, 12 h, 14 h, 20 h and 24 h (on day 1, 2 and 14).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part II
Number analyzed (Participants) | 17
ng/mL
  Midazolam (alone) | 12.24 (4.091)
  Midazolam (co-admin) Day 2 | 13.69 (5.892)
  Midazolam (co-admin) Day 14 | 13.53 (6.092)

ADVERSE EVENTS:
Time Frame: Period I, Part I: AEs (including SAEs) were collected from start of IMP administration (Day 1) until the end-of-study visit on Day 14. Period II, Part II: AEs (including SAEs) were collected from start of IMP administration (Day 1) until the end-of-study visit on Day 22.
Description: The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0. AEs were assessed as unlikely, possibly, or probably related to the IMPs.
Arm/Group | Part I | Part II
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 11/17 | 8/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I (N=17) | Part II (N=18)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05633147/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT05633147/SAP_001.pdf